CLINICAL TRIAL: NCT07151144
Title: The Impact of Massage and Shower, as Non-Pharmacological Interventions During Labor, on Birth Satisfaction, Maternal Comfort, and Breastfeeding Success
Brief Title: Effects of Massage and Shower on Birth Experience and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Eda Gökmen
Record Dates: First submitted 2025-07-18; First posted 2025-09-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy; Delivery Care
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Massage and Showe
  Interventions: Other: Massage; Other: Shower
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Massage — During the active phase of labor (cervical dilation of 4-7 cm), participants received 15-minute sessions of light-pressure massage to the lower back, sacrum, and lumbar area at regular intervals.
  Arms: intervention group
Other: Shower — During the same phase, participants were assisted to take a warm shower for approximately 20 minutes.
  Arms: intervention group

SUMMARY:
Study Design This study is a quasi-experimental research designed to examine the effects of massage and warm shower-used as non-pharmacological methods during labor-on birth satisfaction, maternal comfort, and breastfeeding success.

tudy Population

The study was conducted in the delivery unit of a public hospital in Turkey in 2025. The sample consisted of women who were experiencing their first pregnancy and giving birth for the first time. Inclusion criteria were as follows:

Between 37 and 42 weeks of gestation,

Low-risk, singleton pregnancies,

Planned for vaginal delivery,

No significant obstetric complications during pregnancy,

Voluntarily agreed to participate in the study.

A total of 120 participants were randomly assigned into three groups:

Massage Group (n=430): Received massage during labor.

Shower Group (n=40): Took a warm shower during labor.

Control Group (n=40): Received routine standard hospital care without any additional intervention.

Data Collection Tools

Data were collected using the following instruments:

Personal Information Form

Birth Satisfaction Scale

Birth Comfort Scale

Breastfeeding Success Scale Intervention Massage Group: During the active phase of labor (cervical dilation of 4-7 cm), participants received 15-minute sessions of light-pressure massage to the lower back, sacrum, and lumbar area at regular intervals.

Shower Group: During the same phase, participants were assisted to take a warm shower for approximately 20 minutes.

Control Group: Received routine intrapartum care with no additional non-pharmacological intervention

DETAILED DESCRIPTION:
Before the intervention (baseline during early labor),

Immediately after birth (for comfort and satisfaction),

Within the first 2 hours postpartum (for breastfeeding success).

ELIGIBILITY:
Inclusion Criteria:

Between 37 and 42 weeks of gestation,

Low-risk, singleton pregnancies,

Planned for vaginal delivery,

No significant obstetric complications during pregnancy,

Voluntarily agreed to participate in the study.

Exclusion Criteria:

-

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Birth Satisfaction | up to 3 months
  Evaluated using the Birth Satisfaction Scale (BSS), which measures a mother's satisfaction with her labor and delivery experience (The scale is a 30-item Likert-type scale. The lowest possible score is 30, and the highest is 150. A higher score indicates higher birth satisfaction.). The scale includes multiple dimensions such as quality of care, personal attributes, and stress experienced during labor.
  25 September, 2025-15 December, 2025
Maternal Comfort | up to 3 months
  Maternal Comfort: Assessed through the Birth Comfort Scale, which evaluates physical, emotional, and environmental aspects of comfort experienced by the mother during labor (The scale is a 34-item Likert-type scale. The lowest possible score is 34, and the highest is 170. A higher score indicates higher postpartum comfort).
  25 September, 2025-15 December, 2025
Breastfeeding Success: | Within the first 2 hours postpartum
  Measured within the first hours postpartum using the LATCH Breastfeeding Assessment Tool, which assesses five components: Latch, Audible swallowing, Type of nipple, Comfort (breast/nipple), and Hold (positioning).A low score indicates unsuccessful breastfeeding, while a high score indicates successful breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethically, patient information can be shared upon reasonable request without revealing their identities for security reasons.